CLINICAL TRIAL: NCT04817839
Title: Optimal Duration of Post-Operative Activity Restriction After Midurethral Sling Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2000029067; 000 (Other: CTGTY)
Record Dates: First submitted 2021-03-23; First posted 2021-03-26 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Urinary Stress Incontinence
Keywords: post-operative physical restrictions
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3-week post-operative activity restriction (Experimental): Participants will be given postoperative instructions which include refraining from lifting anything over 20 pounds, avoiding strenuous exercise, running, or performing high-impact aerobic activities for 3-weeks post operation.
  Interventions: Behavioral: 3-week post-operative activity restriction
- 6-week post-operative activity restriction (Experimental): Participants will be given postoperative instructions which include refraining from lifting anything over 20 pounds, avoiding strenuous exercise, running, or performing high-impact aerobic activities for 6-weeks post operation.
  Interventions: Behavioral: 6-week post-operative activity restriction

INTERVENTIONS:
Behavioral: 3-week post-operative activity restriction — Participants will be given postoperative instructions which include refraining from lifting anything over 20 pounds, avoiding strenuous exercise, running, or performing high-impact aerobic activities for 3-weeks post operation.
  Arms: 3-week post-operative activity restriction
Behavioral: 6-week post-operative activity restriction — Participants will be given postoperative instructions which include refraining from lifting anything over 20 pounds, avoiding strenuous exercise, running, or performing high-impact aerobic activities for 6-weeks post operation.
  Arms: 6-week post-operative activity restriction

SUMMARY:
The purpose of this study is to compare postoperative outcomes and patient satisfaction between 3 and 6-week postoperative restrictions after a midurethral sling procedure.

DETAILED DESCRIPTION:
This is a blinded, randomized controlled trial. Patients undergoing midurethral sling placement for stress urinary incontinence will be asked to participate in the study. If eligible and willing to participate, patients will be randomized to a "3 weeks post-operative restriction" or "6-week post-operative restriction" of activities group.

Currently, pelvic surgeons' recommendations for activity and lifting restrictions during post-operative period vary widely from 1 to 50 pounds (10). Given variation in literature and reasonable expectations for lifting restrictions, 20-pound lifting restriction was considered to be a reasonable and attainable expectation from patients. Both groups will be given an identical set of postoperative instructions which include refrainment from lifting anything over 20 pounds, avoid strenuous exercise, running, or perform high-impact aerobic activities during the restricted activity period. Depending on their random allocation, patients will follow these instructions either for 3 or 6 postoperative weeks. The activities which all patients will be allowed to do during their postoperative recovery include walking, using stairs and showering in both groups. All patient will be asked to refrain from sexual intercourse for 6 weeks consistent with current routine post op recommendations (6). Other than the time of activity restriction post op (heavy lifting, strenuous exercise, running, high impact exercise), patients will receive identical postoperative instructions otherwise.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age,
* Patients who are ambulatory and scheduled for midurethral sling placement surgery only for treatment of stress urinary incontinence

Exclusion Criteria:

* • Patients who are unable to read, understand, or complete study documents in English or Spanish

  * Patient undergoing concomitant surgery for pelvic organ prolapse other than midurethral sling
  * Patients who are unable to commit to 6 weeks of no heavy lifting (20 lbs)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Females only
Enrollment: 206 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2024-12-16 (Actual)

PRIMARY OUTCOMES:
Change in urogenital distress inventory (UDI) stress score | Baseline, 6 Months
  UDI form calculator assesses life quality and symptom distress in women suffering from urinary incontinence. The range is 0 to 70, higher means worse, lowers means better (higher is more symptoms.

SECONDARY OUTCOMES:
Patient Global Impression of Improvement (PGI-I) | 6 months
  The Patient Global Impression of Improvement (PGI-I) is a global index that may be used to rate the response of a condition to a therapy (transition scale). The PGI-I is a transition scale that is a single question asking the patient to rate their urinary tract condition now, as compared with how it was prior to before beginning treatment on a scale from 1 (Very much better) to 7 (Very much worse)
Incontinence Impact Questionnaire Short Form (IIQ-7) | 6 months
  Incontinence Impact Questionnaire (IIQ) short form at 6 months. The IIQ-7 has 7 questions that evaluate quality of life related to urinary symptoms. Item responses are assigned values of 0 for "not at all," 1 for "slightly," 2 for "moderately," and 3 for "greatly." The average score of items responded to is calculated. The average, which ranges from 0 to 3, is multiplied by 33 1/3 to put scores on a scale of 0 to 100. Higher scores indicate worse quality of life .
Change in Patient Satisfaction Post-Operative Questionnaire | 6 weeks, 6 months, and 1 year
  This is a questionnaire that will evaluate patient's satisfaction. Assessed on a 5-point Likert scale with question "How satisfied are you with the result of your incontinence surgery." Range is 0-5. Higher number means more satisfied.
Activity Assessment Scale (AAS) | 3 weeks
  This questionnaire is a 13-item postoperative functional activity scale. The AAS is scored from zero to 100 (higher scores=better activity function).
Change in cough stress test | 6 months, 1 year
  Cough stress test is a clinic evaluation to assess stress urinary incontinence. Positive (leaking of urine w cough) or Negative (no leaking urine w cough)

CONTACTS AND LOCATIONS:
Overall Officials: Oz Harmanli, MD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

REFERENCES:
- [Background] FitzGerald MP, Shisler S, Shott S, Brubaker L. Physical Limitations After Gynecologic Surgery, Journal of Pelvic Surgery: May-June 2001 - Volume 7 - Issue 3 - p 136-139